CLINICAL TRIAL: NCT01906151
Title: A Prospective, Open Label Study Assessing the 24-hour Intraocular Pressure Pattern Monitored by SENSIMED Triggerfish® in Primary Angle Closure and Primary Angle Closure Glaucoma Patients, Before and After Laser Peripheral Iridotomy
Brief Title: IOP Pattern in Primary Angle Closure and Primary Angle Closure Glaucoma Patients, Before and After LPI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Sensimed AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TF-1306
Record Dates: First submitted 2013-07-19; First posted 2013-07-23 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SENSIMED Triggerfish® (Other): SENSIMED Triggerfish® (TF) is a CE-marked portable device that monitors the 24-hour intraocular pressure (IOP) pattern by a wireless contact lens sensor (CLS) placed on the eye that sends its signals wirelessly via a periorbital patched adhesive antenna to a recorder. Upon completion, the recording can be transmitted to a computer for read-out and visualization
  Interventions: Device: SENSIMED Triggerfish®

INTERVENTIONS:
Device: SENSIMED Triggerfish® — SENSIMED Triggerfish® (TF) is a CE-marked portable device that monitors the 24-hour intraocular pressure (IOP) pattern by a wireless contact lens sensor (CLS) placed on the eye that sends its signals wirelessly via a periorbital patched adhesive antenna to a recorder. Upon completion, the recording can be transmitted to a computer for read-out and visualization

SUMMARY:
The purpose of the study is to determine the relationship of the intraocular pressure patterns recorded during 2 sessions using Triggerfish, before and after elective laser peripheral iridotomy in angle closure glaucoma patients

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Primary Angle Closure (PAC) or Primary Angle Closure Glaucoma (PACG) with indication for Laser Peripheral Iridotomy (LPI). PAC is defined by the presence of a partial or complete iridotrabecular contact(ITC) in more than 2 quadrants with either raised intraocular pressure (IOP) (ie. more than 21 mmHg) and/or PAS; however, with normal optic disc and visual field. PACG is defined by the presence of ITC with either raised IOP and/or PAS, and evidence of glaucomatous optic disc and visual field
* No IOP-lowering drug treatment or a 4-week wash-out period prior to Study Day 0
* Aged ≥18 years, of either sex
* Not more than 6 diopters spherical equivalent on the study eye
* Have given written informed consent, prior to any investigational procedures

Exclusion Criteria:

* History of acute angle closure glaucoma on the study eye
* Secondary angle closure glaucoma on the study eye
* History of ocular surgery within the last 3 months on the study eye
* History of ocular laser treatment, including previous LPI on the study eye
* Corneal or conjunctival abnormality precluding contact lens adaptation on the study eye
* Severe dry eye syndrome on the study eye
* Patients with allergy to corneal anesthetic
* Patients with contraindications for silicone contact lens wear
* Patients not able to understand the character and individual consequences of the investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the differences between the nycthemeral intraocular pressure patterns recorded with Triggerfish during two 24-hour periods, in patients with Primary angle closure and Primary angle closure glaucoma, before and after laser peripheral iridotomy | 24 hours

SECONDARY OUTCOMES:
To assess the nycthemeral intraocular pressure patterns specific to primary angle closure and primary angle closure glaucoma | 24 hours
To assess the effect of laser peripheral iridotomy on diurnal and nocturnal intraocular pressure pattern in primary angle closure and primary angle closure glaucoma | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Baudouin, MD, Principal Investigator — CHNO des Quinze-Vingts, 28 rue Charenton, 75571 Paris Cedex 12, France
Locations (1):
- CHNO des Quinze-Vingts, 28 rue Charenton, Paris, France